CLINICAL TRIAL: NCT05085678
Title: Development and Evaluation of a PROMs-based Interactive Programme as a Supporting Tool for Breast Cancer Patients Using Adjuvant Endocrine Therapy
Brief Title: Co'Moon for Supporting Breast Cancer Patients on Adjuvant Endocrine Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: G0F9119N
Record Dates: First submitted 2021-08-13; First posted 2021-10-20 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Quality of Life; Self Efficacy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with convenience sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Standard of care:
  * a short overview of the physician on adjuvant endocrine therapy
  * a brochure on adjuvant endocrine therapy
  * a voluntary group session on adjuvant endocrine therapy
  and a monthly questionnaire on the patient reported outcomes
- Intervention group (Experimental): Standard care with the access of to the online tool Co'moon and a monthly questionnaire on patient reported outcomes.
  The outcome of the questionnaires are summarized for the physician to discuss during the follow-up consultation.
  Interventions: Device: Co'moon (online website to support women with AET)

INTERVENTIONS:
Device: Co'moon (online website to support women with AET) — The tool contains three parts:
  1. e-learning based on the brochure on adjuvant endocrine therapy (AET) in the University Hospital Leuven,
  2. serious game where patients are confronted with scenes of their daily life and motivational guidelines to stimulate their self-management,
  3. a patient-reported-outcome questionnaire (PROMs), reported in the patient medical file.
  The tool is designed to stimulate patients self-management of their menopausal AET-related complaints and to discuss them with their health care professionals .
  Other Names: Class 1 medical device
  Arms: Intervention group

SUMMARY:
The objective of the study is to evaluate the effect of an online tool, based on patient reported outcomes (Co'moon), on the quality of life of breast cancer patients on adjuvant endocrine therapy in the University Hospital Leuven.

DETAILED DESCRIPTION:
The project aims to develop and evaluate an online programme to support patients with breast cancer on adjuvant endocrine therapy in the University Hospital Leuven. The tool "Co'moon" has been developed in the first phase of the project and secondly refine in a pilot study. In the third phase a randomised controlled study investigates the effect of Co'moon in comparison with the standard of care in the University Hospital Leuven. Hereby focussing on the improvement of self-efficacy en quality of life.

ELIGIBILITY:
Inclusion Criteria patients:

* Women
* Older than 18 years
* Speaking, understanding and writing Dutch fluently
* Mentally competent
* Recently underwent a operation for breast cancer (invasive or in situ)
* Takes AET for maximum two months
* Consultation planned within 4-5 month
* Home access of a computer with internet connection

Exclusion Criteria patients:

* Different treatments regimes (e.g. adjuvant trial or a combination with cycline-dependent kinase (CDK) 4/6-inhibitors)
* Metastatic disease

Inclusion Criteria health care professionals:

* Contact with patient(s) included in the trial

Exclusion Criteria health care professionals:

* Included in panels
* Member of the research team

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in quality of Life - FACT-ES - B5 - H18 | monthly after two months of AET; up to 3 months
  Total score of Functional Assessment of Chronic Illness Therapy system of Quality of Life questionnaires of endocrine symptoms (FACT-ES) combined with additional questions B5 and H18. A validated questionnaire with a 5-point Likert scale and a total score of 180 (high QoL).
Change in self-efficacy | month 3 and 6 or 7 after the start with AET
  patient reported impact on the side effects of AET
Therapy adherence | monthly after two months of AET; up to 3 months
  patient reported intentional or accidental forgot the medication
Questionnaire on patients experience with the patient-physician relationship | month 6 or 7 after the start with AET
  patient reported their experience of the follow-up consultation in a 5 point Likert scale questionnaire
Questionnaire on change in patient-relative communication over a period of +/- 3 months | month 3 and 6 or 7 after the start with AET
  patient reported a change in the communication of patients with their relatives in a 5 point Likert scale questionnaire

SECONDARY OUTCOMES:
Patient reported outcomes | Monthly after two months of AET; up to 3 months
  Subscales of FACT-ES combined with additional questions B5 and H18.
Questionnaire on the experience of the healthcare professional regarding the summary of PRO's | month 6 or 7 after the start of AET
  the experience of healthcare professionals with the consultation with a 5 point Likert scale questionnaire (1 = strongly disagree, and 5 = strongly agree). The maximum score is 25.
Time-spend on Co'moon | up to 3 months
  Logging of the time women spend on Co'moon

CONTACTS AND LOCATIONS:
Overall Officials: Ines Nevelsteen, Phd, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven campus Gasthuisberg, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No